CLINICAL TRIAL: NCT05135260
Title: The Effects of Virtual Reality on Pain, Stress, and Affect in the Infusion Clinic
Brief Title: Virtual Reality on Pain, Stress, and Affect in the Infusion Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cody Stansel (Other)
Responsible Party: Sponsor-Investigator, Cody Stansel, Principal Investigator, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VICC SUPP 2079
Record Dates: First submitted 2021-11-09; First posted 2021-11-26 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms | interventions — Virtual Reality Exposure Therapy; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Therapy (Experimental): Participants will watch videos for 11 minutes that will allow them to view nature, dinosaurs, animals, and human interactions in three dimension.
  Interventions: Behavioral: Virtual reality therapy; Behavioral: Questionnaires; Procedure: Measure heart rate; Behavioral: Cyber sickness measurement
- Control Group (Active Comparator): This group will not watch videos, but will continue with their normal routine as if nothing has changed.
  Interventions: Behavioral: Questionnaires; Procedure: Measure heart rate

INTERVENTIONS:
Behavioral: Virtual reality therapy — Participants will watch a video allowing them to view nature, dinosaurs, animals, and human interactions in three dimensions during a session lasting 11 minutes.
  Arms: Virtual Reality Therapy
Behavioral: Questionnaires — Questionnaires will be completed regarding stress, pain and affect
Procedure: Measure heart rate — To be measured prior to starting treatment and halfway through the 11 minute Video
Behavioral: Cyber sickness measurement — To be measured using the fast motion sickness scale
  Arms: Virtual Reality Therapy

SUMMARY:
This study will investigate the ability of virtual reality to function as a novel distraction intervention and improve the experience of patients who are receiving chemotherapy in the infusion clinic.

DETAILED DESCRIPTION:
Objectives:

Primary Objective:

- To deploy and evaluate virtual reality as an intervention for stress, pain, and negative affect

Secondary Objective:

- To evaluate cyber sickness and patient satisfaction related to the virtual reality treatment

ELIGIBILITY:
Inclusion Criteria:

* At or above the age of 18
* English Speaking
* Diagnosed with cancer
* No previous history of seizures, losses of awareness, or other symptoms linked to an epileptic condition
* Not sensitive to motion sickness
* Not currently experiencing any contagious conditions, infections, or diseases (particularly of the eyes, skin, or scalp)
* Does not use a device to regulate heart rate or rhythm (such as a pacemaker)
* Not taking antiarrhythmic medications
* Not actively receiving radiopharmaceutical therapy

Exclusion:

* To ensure that there is sufficient time to complete the virtual reality treatment, patients who are scheduled for visits for periods of less than one hour will not be included in this study. Additionally, patients must consent to participating in the study on the day of the experience.
* Patients who are asleep prior to consenting will not be asked to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Positive or negative effect of Virtual Reality therapy on improving the experience of participants receiving chemotherapy | Approximately 12 months
  Measured by the Positive and Negative Affect Scale (0=minimum to 5=maximum). Consisting of a number of words that describe different feelings and emotions. Patients are instructed to indicate to what extent they currently feel each of the feelings or emotions. Afterwards, patient responses are scored to produce a numerical positive affect score and a negative affect score.
Measure the affect of Virtual Reality Therapy on improving stress | Approximately 12 months
  Measured by stress level using the stress numerical rating
Measure the affect of Virtual Reality Therapy on improving pain | Approximately 12 months
  Measured by pain level using the pain numerical score (scale 0 (none) to 10 (worst)

SECONDARY OUTCOMES:
Rate of cyber sickness (Virtual Reality Therapy Arm Only) | Approximately 12 months
  Measured with the Fast MS Scale (FMS), a verbal rating scale ranging from zero (no sickness at all) to 20 (frank sickness).

CONTACTS AND LOCATIONS:
Overall Officials: Cody Stansel, MSN, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT05135260/ICF_000.pdf